CLINICAL TRIAL: NCT01027923
Title: A Phase I Study of Intravenous Plerixafor in Combination With Mitoxantrone Etoposide and Cytarabine for Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: IV Plerixafor With Mitoxantrone Etoposide and Cytarabine for Acute Myeloid Leukemia (AML)
Acronym: AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawal of support from sponsor
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-1825 / 201101703
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — plerixafor; Mitoxantrone; Etoposide; etoposide phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level 1 (Experimental): Mitoxantrone 8 mg/m2/day IV over 30 minutes once daily on days 1-5
  Plerixafor 320 mcg/kg/day IV over 30 minutes on days 0-5
  Etoposide 100 mg/m2/day IV over 60 minutes once daily on days 1-5
  Cytarabine 1000 mg/m2/day IV over 60 minutes once daily on days 1-5
  Interventions: Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Dose Level 2 (Experimental): Mitoxantrone 8 mg/m2/day IV over 30 minutes once daily on days 1-5
  Plerixafor 420 mcg/kg/day IV over 30 minutes on days 0-5
  Etoposide 100 mg/m2/day IV over 60 minutes once daily on days 1-5
  Cytarabine 1000 mg/m2/day IV over 60 minutes once daily on days 1-5
  Interventions: Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine
- Dose Level 3 (Experimental): Mitoxantrone 8 mg/m2/day IV over 30 minutes once daily on days 1-5
  Plerixafor 560 mcg/kg/day IV over 30 minutes on days 0-5
  Etoposide 100 mg/m2/day IV over 60 minutes once daily on days 1-5
  Cytarabine 1000 mg/m2/day IV over 60 minutes once daily on days 1-5
  Interventions: Drug: Plerixafor; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: Plerixafor
  Other Names: AMD3100; Mozobil
Drug: Mitoxantrone
  Other Names: Novantrone
Drug: Etoposide
  Other Names: Etopophos; Toposar; VePesid; VP156
Drug: Cytarabine
  Other Names: Cytosar-U; Ara-C; Cytosine arabinoside

SUMMARY:
In this phase I extension study, the investigators seek to test the safety of both higher doses of plerixafor as well as intravenous dosing to maximize inhibition of the target, CXCR4.

DETAILED DESCRIPTION:
In this study, we are seeking to target the leukemia microenvironment to overcome disease resistance. We hypothesize that by disrupting the interaction of leukemic blasts with the bone marrow microenvironment, we may sensitize leukemic blasts to the effects of cytotoxic chemotherapy. In current formulations, the volume of plerixafor required to administer doses higher than 240 mcg/kg may result in significant discomfort with repeated daily injections. In this phase I extension study, we seek to test the safety of both higher doses of plerixafor as well as intravenous dosing to maximize inhibition of the target, CXCR4.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia diagnosed according to WHO criteria with one of the following:

  * Primary refractory disease following ≥ 1 round of induction chemotherapy
  * First relapse or higher
* Age between 18 and 70 years
* ECOG performance status ≤ 2
* Adequate organ function defined as:

  * Creatinine ≤ 1.5 x institutional ULN
  * AST ≤ 2 x ULN except when in the opinion of treating physician is due to direct involvement of leukemia (e.g., hepatic infiltration or biliary obstruction due to leukemia)
  * ALT ≤ 2 x ULN except when in the opinion of treating physician is due to direct involvement of leukemia (e.g., hepatic infiltration or biliary obstruction due to leukemia)
  * Total bilirubin ≤ 2 x ULN except when in the opinion of treating physician is due to direct involvement of leukemia (e.g., hepatic infiltration or biliary obstruction due to leukemia)
  * Left ventricular ejection fraction of ≥ 40% by MUGA scan or echocardiogram
* Women of childbearing potential and sexually active males must be willing and able to use effective contraception while on study
* Able to provide signed informed consent prior to registration on study

Exclusion Criteria:

* Acute promyelocytic leukemia (AML with t(15;17)(q22;q11) and variants)
* Peripheral blood blast count ≥ 50 x 103 /mm3
* Active CNS involvement with leukemia
* Previous treatment with MEC or other regimen containing both mitoxantrone and etoposide
* Pregnant or nursing
* Concurrently receiving any other investigational agent
* Received colony stimulating factors filgrastim or sargramostim within 48 hours or pegfilgrastim within 14 days of study
* Less than 2 weeks from the completion of any previous cytotoxic chemotherapy (excluding hydroxyurea)
* Severe concurrent illness that would limit compliance with study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and dose limiting toxicities of intravenous plerixafor when combined with MEC in patients with relapsed or refractory AML. | Days 1-42 (all patients have to complete)

SECONDARY OUTCOMES:
To determine the complete response rate (CR) for plerixafor when combined with MEC in patients with relapsed or refractory AML. | Between days 15-42
To determine the safety and tolerability of plerixafor in combination with MEC | Minimum of 30 days following completion of treatment
To determine the PK and explore potential PK drug-drug interactions between plerixafor and MEC. | Predose, 15 min, 30 min , and 10 hrs
To determine the time to hematologic recovery | For up to 2 years
To characterize the mobilization of leukemic cells with plerixafor plus G-CSF. | Baseline, 6 hours
To characterize the effects of plerixafor plus G-CSF on SDF-1/CXCR4 signaling on leukemic blasts. | Baseline, 6 hours
To determine the time to overall survival | For up to 2 years
To determine the time to event-free survival | For up to 2 years
To determine the time to duration of remission | For up to 2 years
To determine the time to relapse-free survival | For up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Uy, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu